CLINICAL TRIAL: NCT05248841
Title: A Single Center, Single-dose, Double-blind, Randomized, Two-period, Two-treatment, Two-sequence, Crossover Study to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity Between HEC-Glargine and US-Lantus® Using the Euglycemic Clamp Technique in Healthy Male Adult Volunteers
Brief Title: A Study to Demonstrate Pharmacokinetic and Pharmacodynamic Biosimilarity Between HEC-Glargine and US-Lantus® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lannett Company, Inc. (Industry)
Collaborators: Parexel (Industry); FARMOVS (Pty) Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LC-INS-2001; PIND147873 (Other: USFDA Identifying Number)
Record Dates: First submitted 2022-01-24; First posted 2022-02-21 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: pharmacokinetic; pharmacodynamic; euglycemic clamp technique; insulin glargine; biosimilarity study
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HEC-Glargine Treatment A (Test) (Experimental): Subjects will receive single doses of Test Formulation HEC-Glargine on Day 1 of Treatment periods 1 and 2 followed by at least 7-21 days washout.
  Interventions: Drug: HEC-Glargine
- US-Lantus Treatment B (Reference) (Active Comparator): Subjects will receive single doses of Reference Formulation Lantus on Day 1 followed of Treatment periods 1 and 2 by at least 7-21 days washout.
  Interventions: Drug: US-Lantus

INTERVENTIONS:
Drug: HEC-Glargine — Subjects will receive 0.5 IU/kg of HEC-Glargine subcutaneously as a single morning dose on Day 1.
  Arms: HEC-Glargine Treatment A (Test)
Drug: US-Lantus — Subjects will receive 0.5 IU/kg of Lantus subcutaneously as a single morning dose on Day 1.
  Other Names: Insulin glargine
  Arms: US-Lantus Treatment B (Reference)

SUMMARY:
This is a phase 1 study to demonstrate pharmacokinetic and pharmacodynamic similarity between HEC-Glargine and US-Lantus® using the euglycemic clamp technique in healthy male adult volunteers.

DETAILED DESCRIPTION:
This will be a double-blind, single-dose, randomized, two-period, two-treatment, two-sequence crossover clamp study performed at a single study center. The study population consists of healthy adult male subjects.

The study will comprise of:

* A screening period: maximum 28 days prior to first dose administration.
* Admission: Subjects will be admitted to the study center on Day -1
* Two Treatment Periods (Treatment Periods 1 and 2): Subjects will be randomized to either of the 2 treatment sequences (AB or BA) on Day 1 of Treatment Period 1 to receive either test or reference product as per randomization schedule in a 1:1 ratio.

  * Treatment A (Test Formulation): HEC-Glargine
  * Treatment B (Reference Formulation): US-Lantus®

On Day 1 of each Treatment Period, the study drug or reference product will be administered as a single morning dose to subjects in a fasting state. There will be a wash-out period of at least 7 calendar days. Each subject will receive both test and reference products in a crossover pattern over Treatment Periods 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Participant has body weight not less than 60 kg and body mass index between 18.5 and 30.0 kg/m^2 (both inclusive).
* Glycohemoglobin (HbA1c) levels are <6.0%.
* Normal oral glucose tolerance test conducted within the previous 6 months
* Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations should be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests
* Non-smokers or mild to moderate smokers (≤ 10 cigarettes or pipes per day).

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use >21 units of alcohol per week
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter or herbal remedies
* Participation in another study with an experimental drug, where the last administration of the previous study drug was within 12 weeks before administration of study drug in this study.
* Treatment within the previous 3 months before the first administration of study drug with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major disease (i.e., a disease that could not be treated at home, but the subject had to be hospitalized or needed general anesthesia usually for a major operation) during the 3 months before commencement of the screening period.
* Positive test for insulin antibodies.
* History of bronchial asthma or any other bronchospastic disease, and/or convulsions, and/or porphyria.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Resting pulse of >100 beats per minute (bpm) or <40 bpm during the screening period, either supine or standing.
* Hypertension diagnosed during screening or current diagnosis of hypertension.
* Hemoglobin count deviating more than 10% of the lower limit of normal.
* Clinically relevant abnormalities in the coagulation status.
* History of bleeding disorders.
* Veins unsuitable for venous blood collection and cannulation.
* Any specific study drug safety concern.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 104 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from 0 hours to 24 hours (AUC0-24h) of M1 | Day 1 and Day 2
  The Pharmacokinetics (PK) parameters of HEC-Glargine to the US-approved Lantus® insulin glargine injection (US-Lantus®) solution for SC injection to demonstrate PK similarity for insulin glargine and/or metabolite 21A-Gly-human insulin (M1) will be assessed.
Maximum observed plasma exogenous insulin glargine concentration (Cmax) of M1 | Day 1 and Day 2
  The PK parameters of HEC-Glargine to the US-approved Lantus® insulin glargine injection (US-Lantus®) solution for SC injection to demonstrate PK similarity for insulin glargine and/or metabolite 21A-Gly-human insulin (M1) will be assessed.
Area under the Glucose infusion rate (GIR) -time curve (calculated as the exact area under the stepwise constant function) from 0 hours to 24 hours (GIRAUC0-24h) | Day 1 and Day 2
  The pharmacodynamics (PD) of HEC-Glargine to US-Lantus®, by means of GIR profiles after single SC dose will be assessed.
Maximum GIR (GIRmax) | Day 1 and Day 2
  The PD of HEC-Glargine to US-Lantus®, by means of GIR profiles after single SC dose will be assessed.

SECONDARY OUTCOMES:
Area under the concentration-time curve from 0 hours to the last quantifiable concentration-time (AUC0-t) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed. Also, AUC0-t will be evaluating the inter-subject and intra-subject variability of PK of HEC-Glargine in comparison to US-Lantus®, assessed by intra-subject coefficients of variation for primary PK parameters.
Area under the concentration-time curve from 0 hours to 6 hours (AUC0-6h) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the concentration-time curve from 6 hours to 12 hours (AUC6-12h) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the concentration-time curve from 0 hours to 12 hours (AUC0-12h) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the concentration-time curve from 12 hours to 18 hours (AUC12-18h) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the concentration-time curve from 18 hours to 24 hours (AUC18-24h) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the concentration-time curve from 12 hours to 24 hours (AUC12-24h) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Time to maximum plasma exogenous insulin glargine concentration (Tmax) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the concentration-time curve from 0 hours to the last quantifiable concentration-time extrapolated to infinity (AUC0-∞) | Day 1 and Day 2
  The PK parameters of HEC-Glargine, US-Lantus®, and M1 will be assessed.
Area under the GIR-time curve for the time of a dosing interval (GIRAU0-t) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed. Also, GIRAU0-t will be evaluating the inter-subject and intra-subject variability of PD of HEC-Glargine in comparison to US-Lantus®, assessed by intra-subject coefficients of variation for primary PD parameters.
Area under the GIR-time curve from 0 hours to end of clamp (GIRAUC0-end of clamp) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 0 hours to the last quantifiable concentration-time with extrapolation to infinity (GIRAUC0-∞) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 0 hours to 6 hours (GIRAUC0-6h) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 6 hours to 12 hours (GIRAUC6-12h) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 0 hours to 12 hours (GIRAUC0-12h) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 12 hours to18 hours (GIRAUC12-18h) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 18 hours to 24 hours (GIRAUC18-24h) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Area under the GIR-time curve from 12 hours to 24 hours (GIRAUC12-24h) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Time to maximum glucose infusion rate (TGIRmax) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Total amount of glucose infused during clamp procedure (Gtot) | Day 1 and Day 2
  The PD parameters of HEC-Glargine, US-Lantus® will be assessed.
Time to onset of action (TOA) | Day 1 and Day 2
  The TOA will be assessed for HEC-Glargine, US-Lantus® as PD parameters.
Maximum observed plasma exogenous insulin glargine concentration (Cmax) | Day 1 and Day 2
  The Cmax will be evaluating the inter-subject and intra-subject variability of PK of HEC-Glargine in comparison to US-Lantus®, assessed by intra-subject coefficients of variation for primary PK parameters.
Maximum GIR (GIRmax) | Day 1 and Day 2
  The GIRmax will be evaluating the inter-subject and intra-subject variability of PD of HEC-Glargine in comparison to US-Lantus®, assessed by intra-subject coefficients of variation for primary PD parameters.
Number of subjects with adverse events (AEs) | Day -1 to within 7 Days of completion of the last period or early withdrawal (approximately 31 days)
  To assess safety and tolerability of the HEC-Glargine compared to US-Lantus® after single SC dose To assess safety and tolerability of the HEC-Glargine compared to US-Lantus® after single SC dose

CONTACTS AND LOCATIONS:
Locations (1):
- FARMOVS Clinical Research Organization, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: Undecided